CLINICAL TRIAL: NCT00871247
Title: Randomized, 2-Way Crossover Bioequivalence Study Finasteride 5 mg Tablet and Proscar Administrated as 1 x 5 mg Tablet in Healthy Subjects Under Fed Conditions
Brief Title: A Relative Bioavailability Study of Finasteride 5 mg Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Meena Venugopal, Director, Clinical R&D, Actavis Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 40398
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Bioequivalence; finasteride; Healthy subjects
MeSH Terms: interventions — Finasteride; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Finasteride 5 mg single dose tablet, single dose
  Interventions: Drug: Finasteride 5 mg Tablet, single dose
- B (Active Comparator): Proscar® 5 mg Tablet, single dose
  Interventions: Drug: Proscar® 5 mg Tablet, single dose

INTERVENTIONS:
Drug: Finasteride 5 mg Tablet, single dose — A: Experimental Subjects received Intas Pharmaceuticals Ltd, India formulated products under fed conditions
  Other Names: Finasteride
  Arms: A
Drug: Proscar® 5 mg Tablet, single dose — B: Active comparator Subjects received Merck Sharp and Dohme, U.S.A formulated products under fed conditions
  Other Names: Finasteride
  Arms: B

SUMMARY:
The purpose of this study is to compare the rate and extent of absorption of Actavis Group hf, Iceland, finasteride and Merck & Co. Inc., U.S.A. (Proscar), finasteride, administered as a 1 x 5 mg tablet, under fed conditions.

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: Randomized, 2-period, 2-sequence, crossover design.

Official Title: Randomized, 2-Way Crossover, Bioequivalence Study of Finasteride 5 mg Tablet and Proscar Administered as 1 x 5 mg Tablet in Healthy Subjects Under Fed Conditions

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

Rate and Extend of Absorption

ELIGIBILITY:
Inclusion Criteria:

* Male, smoker or non-smoker, 18 years of age and older.
* Capable of consent.
* BMI ~19.0 and <30.0 kg/m2 Sexual abstinence for the duration of the study is recommended given the potential harm to a fetus from migration of this drug to the semen. Sexually-active males must refrain from heterosexual intercourse without the use of a condom for a period of one week from the initial dosing.

Exclusion Criteria:

* Clinically significant illnesses within 4 weeks prior to the administration of the study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any clinically significant abnormality found during medical screening.
* Any reason which, in the opinion of the Medical Sub-Investigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive testing for hepatitis B, hepatitis C, or HN at screening.
* EeG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
* History of significant alcohol abuse or drug abuse within one year prior to the screening visit.
* Regular use of alcohol within six months prior to the screening visit (more than fourteen units of alcohol per week [I Unit:= 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).
* Use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP] and crack) within 1 year prior to the screening visit or positive urine drug screen at screening.
* History of allergic reactions to heparin, finasteride, or other related drugs.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; examples of inhibitors: antidepressants (SSRI), cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluoroquinolones, antihistamines) within 30 days prior to administration of the study medication.
* Use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication .
* Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug.
* Any clinically significant history or presence of clinically significant neurological, endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric, or metabolic disease.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (incl~ding natural food supplements, vitamins, garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Difficulty to swallow study medication.
* Smoking more than 25 cigarettes per day.
* Any food alIergy, intolerance, restriction or special diet that, in the opinion of the Medical Sub-Investigator, could contraindicate the subject's participation in this study.
* A depot injection or an implant of any drug within 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 7 days prior to drug administration. Donation or loss of whole blood (excluding the volume of blood that will be drawn during the screening procedures of this study) prior to administration of the study medication as follows:
* 50 mL to 300 mL of whole blood within 30 days,
* 301 mL to 500 mL of whole blood within 45 days, or
* more than 500 mL of whole blood within 56 days prior to drug administration.
* Consumption of food or beverages containing grapefruit (e.g. fresh, canned, or frozen) within 7 days prior to administration of the study medication.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-11; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Girard, M.D., Principal Investigator — SFBC Anapharm
Locations (1):
- SFBC Anapharm, Sainte-Foy, Quebec, Canada